CLINICAL TRIAL: NCT04802213
Title: Invention of Portable Laser Acupuncture and Joint Mobilization Device on Frozen Shoulder and Therapeutic Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, LJ Hwu, Attending physician, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSMUH-17084
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rehabilitation exercise (Active Comparator): 1.perform rehabilitation exercise for patients with frozen shoulders (10 repetitions of each exercise, three times a day, 3 days a week for 8 weeks)
  Interventions: Other: Rehabilitation exercise
- Rehabilitation exercise + joint mobilization device treatment (Experimental): 1. perform rehabilitation exercise for patients with frozen shoulders (10 repetitions of each exercise, three times a day, 3 days a week for 8 weeks)
  2. perform joint mobilization device treatment for patients with frozen shoulders (The treatment time was total of 30 minutes. Three times a week for 8 continuous weeks.)
  Interventions: Other: Rehabilitation exercise; Device: joint mobilization device treatment
- Rehabilitation exercise +joint mobilization device treatment + laser acupuncture device treatment (Experimental): 1. perform rehabilitation exercise for patients with frozen shoulders (10 repetitions of each exercise, three times a day, 3 days a week for 8 weeks)
  2. perform joint mobilization device treatment for patients with frozen shoulders (The treatment time was total of 30 minutes. Three times a week for 8 continuous weeks.)
  3. perform laser acupuncture device treatment for patients with frozen shoulders ( three sessions per week for 8 consecutive weeks. patients in each treatment session received laser at a dosage of 4 joules/cm2 for the eight chosen position. )
  Interventions: Other: Rehabilitation exercise; Device: joint mobilization device treatment; Device: laser acupuncture device treatment

INTERVENTIONS:
Other: Rehabilitation exercise — Rehabilitation exercise use the methods that suggested by previous studies including finger wall climbing, pendulum exercise, and arms lifting.
Device: joint mobilization device treatment — The joint mobilization treatment used the mobilization device that developed in this research.It is a device developed by using the design of the vibration force generated by the vibration mechanism and the technologies to simulate the mobilization of the shoulder joint.When the subject uses the device, first sit on a seat that can be adjusted according to the user's body shape and buckle the shoulder fixation device. Then use the specially designed shoulder movement setting mechanism of the device to set the user's shoulder movement and movement angle.The next step is to set the direction and magnitude of the vibration force applied by the device to the shoulder joint in accordance with the joint mobilization technique (posterior, anterior, and inferior) that the therapist or user intends to perform to achieve the effect of simulating joint mobilization and increasing joint mobility.
  Arms: Rehabilitation exercise + joint mobilization device treatment; Rehabilitation exercise +joint mobilization device treatment + laser acupuncture device treatment
Device: laser acupuncture device treatment — The laser acupuncture treatment use the laser acupuncture device that developed in this research. A gallium-aluminium-arsenide (GaAlAs, infrared laser) continuous wave diode laser device with a wavelength of 850nm (invisible), a power output of 100 mW, and a spot area of 0.07cm2 was used for laser acupuncture.When performing laser acupuncture treatment, the laser emitted by the device is irradiated on the selected acupuncture points .The acupuncture points (GB 21, LI 4, LI 11, LI 14, LI15, LI 16, SI 9, SI 10, SI 11, TE 14, and TE 15) were determined according to the literature regarding acupuncture application in shoulder pain based on traditional chinese acupuncture.
  Arms: Rehabilitation exercise +joint mobilization device treatment + laser acupuncture device treatment

SUMMARY:
the volunteers with frozen shoulder will be recruited to this experiment and use devices under a designed experimental procedure. After subjects use device , R&D team will collect subject feedback, efficacy assessments, and various device data. This step will not only help investigators to improve and refine the device but also find the best operating mode and using standard of the device to help the frozen shoulder patients.

Subjects in this study will also enter a designed course of treatment. All patients will be distributed equally and randomly to three groups (control , mobilization device, laser acupuncture plus mobilization device) to receive treatment. All groups receive three therapy sessions per week for 8 consecutive weeks. At last, investigators will compare the differences between the three groups to understand the effect of portable laser acupuncture and joint mobilization device on frozen shoulder.

DETAILED DESCRIPTION:
Adhesive capsulitis (also known as frozen shoulder) is a painful and disabling disorder of unclear cause in the shoulder capsule. There are many ways to treat frozen shoulders. Laser acupuncture and joint mobilization are both ways to treat frozen shoulders. According to the literature, laser acupuncture has the effect of pain control for frozen shoulder and joint mobilization can increase the patient's shoulder range of motion. As a creative inspiration, the R&D team uses application and principle of these treatment to design the device. After cooperation and effort, the R&D team developed two devices that are 「portable laser Acupuncture device for frozen shoulder」and「the joint mobilization simulation device」. During the development of two devices, collecting various usage data and user's feelings, feedback and clinical effects are very important. So, R&D team will use this research project to help device development. This project will recruit volunteers as objects for device development and advancement.

The volunteers with frozen shoulder will be recruited to this experiment and use devices under a designed experimental procedure. After subjects use device , R&D team will collect subject feedback, efficacy assessments, and various device data. This step will not only help investigators to improve and refine the device but also find the best operating mode and using standard of the device to help the frozen shoulder patients.

Subjects in this study will also enter a designed course of treatment. All patients will be distributed equally and randomly to three groups (control , mobilization device, laser acupuncture plus mobilization device) to receive treatment. All groups receive three therapy sessions per week for 8 consecutive weeks. At last, investigators will compare the differences between the three groups to understand the effect of portable laser acupuncture and joint mobilization device on frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 25 years old
* Diagnosed with frozen shoulder and pain in the shoulder
* After medical imaging and other related physical examinations, except frozen shoulder, no other shoulder abnormalities and diseases were found.

Exclusion Criteria:

* Suffer from relevant contraindications of this experiment (such as tumor, cancer, etc.);
* Have a history of surgery on the shoulder;
* Have a history of trauma on the shoulder (such as: fracture, dislocation, etc.);
* Suffer from neuromuscular diseases (such as stroke);
* After medical imaging and other related physical examinations, it is found that the shoulder is abnormal and disease other than the frozen shoulder;
* received shoulder steroid injections within 6 months.
* Suffer from contraindications related to the device used in this study.Patients who meet any of the above conditions will be excluded from this experiment.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
shoulder range of motions | 8 consecutive weeks
  shoulder range of motion evaluation, including shoulder flexion, abduction, internal rotation, and external rotation. All shoulder range of motions was measured with a standard goniometer. When measured the shoulder range of motion, the researcher force to the patient's upper limbs to make movements. The endpoint of the movement was where the subject began to feel pain. The therapist stopped applying force and record the degrees of shoulder range of motion.
pain visual analogue scale | 8 consecutive weeks
  pain visual analogue scale that was used to assess levels of pain. The visual analogue scale has been widely used in clinical and research to assess patients with shoulder pain. It is a grading scale from 0cm to 10cm, presented in front of the subject, and the subject selected the location according to their pain during the last 24 hours (0cm indicating "no pain", 10cm indicating "most pain").
disabilities of the arm, shoulder and hand questionnaire | 8 consecutive weeks
  This questionnaire is mainly composed of 30 disability/symptom scales and has been proven to be reliable and effective in evaluating various upper limb dysfunction patients. The scores obtained for all items will be calculated, ranging from 0 (no disability) to 100 (most severely disabled) to evaluate the subject's shoulder condition
constant murley questionnaire | 8 consecutive weeks
  This questionnaire is a tool used to assess the condition of the shoulders. It is a full-point 100-point scale composed of multiple evaluation methods and parameters. The questionnaire is divided into four parts: pain (15 points). activities of daily living (20 points); strength (25 points); and joint mobility (40 points). After completing the questionnaire, add up the scores. The higher the score, the better the shoulder function.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Ting, M.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No